CLINICAL TRIAL: NCT05567458
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Luspatercept (ACE-536) in Chinese Adult Subjects Who Require Regular Red Blood Cell Transfusions Due to Beta (β)-Thalassemia
Brief Title: A Study to Evaluate Luspatercept (ACE-536) in Chinese Participants Who Require Regular Red Blood Cell Transfusions Due to Beta (β)-Thalassemia.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA056-001
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Beta-thalassemia
Keywords: Luspatercept; ACE-536; Transfusion burden
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Luspatercept (Experimental)
  Interventions: Drug: Luspatercept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Luspatercept — Specified dose on specified days
  Other Names: ACE-536; BMS-986346
  Arms: Luspatercept
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of luspatercept plus best supportive care (BSC) versus placebo plus BSC in participants who require regular red blood cell transfusions due to β-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to adhere to the study visit schedule (for example, not scheduled to receive hematopoietic stem cell transplantation [HSCT]) and other protocol requirements.
* Participant has documented diagnosis of β-thalassemia or Hemoglobin E/β-thalassemia (β-thalassemia with mutation and/or multiplication of alpha (α) globin is allowed).
* Participant is regularly transfused, defined as: 6-25 RBC units in the 24 weeks prior to randomization and no transfusion-free period for >42 days during that period.
* Participant has Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.

Exclusion Criteria:

* Participant has a diagnosis of Hemoglobin S/β-thalassemia or α-thalassemia (for example, Hemoglobin H).
* Participant has active hepatitis C virus (HCV) infection as demonstrated by a positive HCVribonucleic acid (RNA) test of sufficient sensitivity, or active infectious hepatitis B virus (HBV) as demonstrated by the presence of hepatitis B surface antigen (HBsAg) and/or HBVdeoxyribonucleic acid (DNA) positive, or known positive human immunodeficiency virus (HIV).
* Participant has a history of deep venous thrombosis or stroke or thromboembolic events (venous or arterial) requiring medical intervention ≤24 weeks prior to randomization.
* Participant uses chronic anticoagulant therapy, unless the treatment stopped at least 28 days prior to randomization. Anticoagulant therapies used for prophylaxis for surgery or high-risk procedures as well as low-molecular-weight heparin for superficial venous thrombosis and chronic aspirin are allowed.
* Participant who has EMH complications requiring treatment to control the growth of EMH mass(es) during the screening period.
* Participant used immunomodulatory imide drugs (IMiDs) ≤ 24 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ≥ 33% reduction from baseline in red blood cell (RBC) transfusion burden over any consecutive 24 weeks | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 - Week 48

SECONDARY OUTCOMES:
Proportion of subjects with ≥ 33% reduction from baseline in RBC transfusion burden during any rolling 24-week interval compared to the 24-week interval prior to start of IP for luspatercept plus BSC versus placebo plus BSC. | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 134
Proportion of participants with ≥ 33% reduction from baseline in RBC transfusion burden over any consecutive 12 weeks | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 134
Proportion of participants with ≥ 50% reduction from baseline in RBC transfusion burden over any consecutive 12 weeks | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 134
Proportion of participants with ≥ 50% reduction from baseline in RBC transfusion burden over any consecutive 24 weeks | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 134
Proportion of participants with ≥ 33% reduction from baseline in RBC transfusion burden over Weeks 13-24 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 13-Week 24
Proportion of participants with ≥ 33% reduction from baseline in RBC transfusion burden over Weeks 37-48 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 37 to Week 48
Proportion of participants with ≥ 33% reduction from baseline in RBC transfusion burden over Weeks 1-24 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 24
Proportion of participants with ≥ 33% reduction from baseline in RBC transfusion burden over Weeks 25-48 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 25 to Week 48
Proportion of participants with ≥ 50% reduction from baseline in RBC transfusion burden over Weeks 13-24 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 13-Week 24
Proportion of participants with ≥ 50% reduction from baseline in RBC transfusion burden over Weeks 37-48 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 37 to Week 48
Proportion of participants with ≥ 50% reduction from baseline in RBC transfusion burden over Weeks 1-24 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 24
Proportion of participants with ≥ 50% reduction from baseline in RBC transfusion burden over Weeks 25-48 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 25 to Week 48
Best change from baseline in total RBC units transfused in 24 weeks within the first 48-week treatment period | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 48
Change from baseline in total RBC units transfused over Weeks 1-24 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 24
Change from baseline in total RBC units transfused over Weeks 25-48 | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 25 to Week 48
Mean change from baseline in serum ferritin | 12 weeks prior to Dose 1 Day 1 (inclusive); Week 37 to Week 48
Change from baseline in Liver Iron Concentration (LIC) (mg/g dw) by magnetic resonance imaging (MRI) | Up to 96 weeks
Change from baseline in myocardial iron by T2-star (T2*) MRI | Up to 96 weeks
Change from baseline in mean daily dose of iron chelation therapy (ICT) | 12 weeks prior to Dose 1 Day 1 (inclusive); Week 37 to Week 48
Change from baseline in self-reported Health-related quality-of-life (HRQoL) assessed by TranQoL | Up to 48 weeks
Change from baseline in self-reported HRQoL assessed by SF-36 | Up to 48 weeks
Proportion of participants who are transfusion independent for any consecutive ≥8 weeks during treatment | Week 1 to Week 134
Proportion of participants who are transfusion independent for any consecutive ≥12 weeks during treatment | Week 1 to Week 134
Duration of reduction in transfusion burden | Week 1 to Week 134
Duration of RBC transfusion independence (TI) | Week 1 to Week 134
Time to response | Week 1 to Week 134
Least number of transfusion events in 24 weeks within the first 48-week treatment period | 24 weeks prior to Dose 1 Day 1 (inclusive); Week 1 to Week 48
Number of participants with Adverse Events (AEs) | Up to 4 years
Frequency of Antidrug antibodies (ADA) | Up to 2 years
Maximum plasma concentration (Cmax) | Up to 2 years
Area under the curve (AUC) | Up to 2 years
Change in spleen volume | Up to 96 weeks
Proportion of subjects, without increase in transfusion burden and with an increase of ≥ 1.0 g/dL in pre-transfusion Hb level on at least 2 separate tests (at least 60 days apart) during any rolling 24-week interval, compared to baseline | 24 weeks prior to Dose 1 Day 1 (inclusive); Dose 1 Day 2 through completion of 48-week treatment for last subject

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- China (10):
  - Local Institution - 0002, Maoming, Guangdong
  - Local Institution - 0005, Shenzhen, Guangdong
  - Local Institution - 0007, Liuchow, Guangxi
  - Local Institution - 0003, Nanning, GX
  - Local Institution - 0006, Haikou, Hainan
  - Local Institution - 0010, Kunming, Yunnan
  - Local Institution - 0009, Guangzhou
  - Local Institution - 0004, Guangzhou
  - Local Institution - 0008, Haikou
  - Local Institution - 0001, Nanning

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html